CLINICAL TRIAL: NCT02852187
Title: Prospective, Randomized, Data Registry Study of MOBIS II Structural Titanium (ST) Interbody Cage Compared to MOBIS Peek Cage for the Treatment of Spondylolisthesis and Degenerative Disc Disease
Brief Title: Single Center Study Comparing MOBIS II ST vs MOBIS PEEK
Acronym: MOBIS_US
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitement
Sponsor: Signus Medizintechnik GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01MOBIS_US
Record Dates: First submitted 2016-07-18; First posted 2016-08-02 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Lumbar Disc Disease
Keywords: Intervertebral Disc Degeneration; Lumbar Spinal Disease
MeSH Terms: conditions — Intervertebral disc disease; Intervertebral Disc Degeneration; Spinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MOBIS PEEK (Active Comparator): Transforaminal Lumbar Interbody Fusion (TLIF) with the SIGNUS MOBIS PEEK Cage
  Interventions: Device: SIGNUS MOBIS PEEK Cage
- MOBIS II ST (Active Comparator): Transforaminal Lumbar Interbody Fusion (TLIF) with the SIGNUS MOBIS II ST Cage
  Interventions: Device: SIGNUS MOBIS II ST Cage

INTERVENTIONS:
Device: SIGNUS MOBIS PEEK Cage — Lumbar Interbody Fusion
  Arms: MOBIS PEEK
Device: SIGNUS MOBIS II ST Cage — Lumbar Interbody Fusion
  Arms: MOBIS II ST

SUMMARY:
Prospective randomized clinical study comparing SIGNUS MOBIS PEEK vs SIGNUS MOBIS II ST in patients with Degenerative Disc Disease at one or two contiguous levels from L2-S1

DETAILED DESCRIPTION:
The protocol includes skeletally mature patients both male and female, 18 to 89 years old, with degenerative disc disease (DDD) at one or two contiguous levels from L2-S1. DDD is defined as discogenic back pain with degeneration of the disc confirmed by patient history and radiographic studies. Patients may also have up to a Grade I spondylolisthesis or retrolisthesis at the involved level(s). Patient should have completed at least six (6) months of non-operative treatment. Patients may have had a previous non-fusion surgery at the involved spinal level(s) and will be followed clinically up to two years.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has symptomatic degenerative disc disease (DDD) at one or two contiguous levels from L2-S1.
2. The patient has documented conservative (non-operative) treatment for at least 6 months.
3. The patient has a VAS back pain of ≥ 60 mm.
4. The patient has an ODI ≥ 40%.
5. The patient is at least 18 years of age and skeletally mature.
6. The general condition of the patient is appropriate for surgery, as evaluated by the Investigator.
7. The patient is willing and able to comply with study requirements.
8. The patient has agreed to participate in the study.

Exclusion Criteria:

1. The patient has undergone any prior spinal fusion surgery at the proposed treatment level(s).
2. The patient has osteoporosis or severe osteopenia as determined by the Investigator. A clinical SCORE calculator may be utilized for females over 40 years of age.
3. The patient has grade 2 or higher spondylolisthesis or retrolisthesis at the affected level(s).
4. The patient has diffuse multilevel neoplastic disease such that no adjacent normal segments exist for engagement or instrumentation.
5. The patient has an active infection.
6. The patient is pregnant or is planning on becoming pregnant in the next two years.
7. The patient is mentally ill or has a history of drug abuse or severe depression/ psychosocial issues.
8. The patient has a known allergy to polyether ether ketone (PEEK), stainless steel or tantalum/titanium.
9. The patient is currently enrolled in an investigational spine study.
10. The patient has rheumatoid arthritis, ankylosing spondylitis or other autoimmune disease.
11. The patient has symptomatic fibrous arachnoiditis

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Fusion rates | 24 Months
  Lumbar fusion demonstrated by radiographic evidence based on plain radiographs, and CT Scans

SECONDARY OUTCOMES:
Subsidence | 24 Months
  disc height demonstrated by radiographic evidence based on plain radiographs, and CT Scans
Patient Reported Outcomes: Visual Analog Scale (VAS) | Through 24 Months
  Comparison of pre-operative to post-operative evaluations
Patient Reported Outcomes: Oswestry Disability Index | Through 24 Months
  Comparison of pre-operative to post-operative evaluations
Patient Reported Outcomes: Evaluations of Quality of Life (QOL) by the EQ-5D-5L | Through 24 Months
  Comparison of pre-operative to post-operative evaluations

CONTACTS AND LOCATIONS:
Overall Officials: William F. Lavelle, MD, Principal Investigator — Upstate Orthopedics
Locations (1):
- Upstate Orthopedics, East Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No